CLINICAL TRIAL: NCT01880827
Title: The Effects of Glucose-dependent Insulinotrophic Peptide (GIP) and Glucagon-like Peptide 1 (GLP-1) on Splanchnic Redistribution of Blood Flow at Postprandial State and After Roux-en-Y Gastric Bypass and Sleeve
Brief Title: Splanchnic Blood Redistribution After Incretin Hormone Infusion and Obesity Surgery
Acronym: GIP-PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Pirjo Nuutila, Professor, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-002689-10
Record Dates: First submitted 2013-02-25; First posted 2013-06-19 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: GIP; GLP-1; type 2 diabetes; obesity; splanchnic blood flow; incretin hormones
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Anastomosis, Roux-en-Y; Glucagon-Like Peptide 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Royx-en-Y surgery (Active Comparator): Mixed meal test (MMS) with flow studies before and 2 months after the operation
  Interventions: Procedure: Roux-en-Y; Drug: GIP-infusion; Drug: MMS
- Control (Active Comparator): Healthy volunteer group, GIP, GLP-1 and MMS studies
  Interventions: Drug: GIP-infusion; Drug: GLP-1; Drug: MMS
- Sleeve gastrectomy (Experimental): Mixed meal test (MMS) with flow studies before and 2 months after the operation
  Interventions: Drug: GIP-infusion; Drug: MMS; Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y — Subjects in the intervention group will be divided into two consecutive surgical groups, RYGB or SG. After the surgery, subjects are controlled in hospital ward for approximately three days.
  Arms: Royx-en-Y surgery
Drug: GIP-infusion — Blood flow and volume during infusion
Drug: GLP-1 — Blood flow and volume during infusion
  Arms: Control
Drug: MMS — Blood flow and volume after meal solution
Procedure: Sleeve gastrectomy — as in RYGS group
  Arms: Sleeve gastrectomy

SUMMARY:
Obesity is a worldwide problem and leads to multiple metabolic and endocrinological problems.

Bariatric surgeries are a growing field as a treatment choice for morbid obesity (BMI > 35 kg/m2). Clinical and research evidence shows that shortly after RYGB, T2DM resolves with improving glucose tolerance. Foregut hypothesis behind bariatric surgeries postulate, that bypassed portions of intestine contain a substance, that acts as an anti-incretin, ie. to counteract metabolically favourable incretins. In view of the recent studies, it may be that GIP is really the anti-incretin behind this hypothesis.

The current study is conducted to investigate the vasoactive roles of the GIP. The investigators aim to show that GIP is the major contributor to the blood flow and tissue blood volume observed in postprandial state.

DETAILED DESCRIPTION:
Obesity is a worldwide problem and leads to multiple metabolic and endocrinological problems, including type 2 diabetes mellitus (T2DM). In T2DM, body is unable to response to circulating insulin levels, which ultimately destroys pancreatic β-cells, leading to chronic hyperglycaemia with ensuing consequences

Intestine is able to produce endocrinologically active substances, which affect to body's intermediary metabolism. One of these substances in glucose-dependent insulinotrophic polypeptide (GIP, part of the incretin family), which potentiates the release of insulin postprandially. However, recent evidence suggests, that GIP may have more harmful than beneficial role in the pathogenesis: it has been shown that GIP participates in the development of insulin resistance, the key defect in the process of metabolic dysfunction. GIP may also regulate postprandial redistribution of splanchnic blood flow which might act in the body's nutrition handling [8].

Bariatric surgeries are a growing field as a treatment choice for morbid obesity (BMI > 35 kg/m2). Most established of these procedures is a Roux-en-Y gastric bypass (RYGB), where duodenum and proximal jejunum is bypassed. Clinical and research evidence shows that shortly (before any significant weight loss) after RYGB, T2DM resolves with improving glucose tolerance. Foregut hypothesis behind bariatric surgeries postulate, that bypassed portions of intestine contain a substance, that acts as an anti-incretin¬, ie. to counteract metabolically favourable incretins. In view of the recent studies, it may be that GIP is really the anti-incretin behind this hypothesis.

Positron emission tomography (PET) is a modern imaging technique, which can be used to study perfusion and metabolism of different organs non-invasively. When radiowater measurement is combined with [15O]CO, both tissues specific perfusion and blood volume can be measured, respectively. When coupled with magnetic imaging (ie. PET-MRI), the volumes-of-interests can be accurately drawn to the desired organs.

The current study is conducted to investigate the vasoactive roles of the GIP. We aim to show that GIP is the major contributor to the blood flow and tissue blood volume observed in postprandial state. Moreover, we hypothesize that the elimination of GIP-effect has a central role in the improved intermediary metabolism observed after bariatric surgery procedures, and that part this change is mediated by changes in splanchnic circulation. Furthermore, we investigate the effect of GLP-1 (glucagon-like peptide 1, another member of incretin family) on splanchnic circulation.

In the present study intestinal, hepatic and pancreatic blood flow and volume are measured using [15O]H2O- and [15O]CO radiotracers and PET-MRI imaging in healthy normal weight volunteers (n = 20, BMI ≤ 27 kg/m2) and in morbidly obese T2DM patients (n = 30, BMI ≤ 35 kg/m2) before and after the bariatric surgery operation. The PET imaging will be performed at fasting state but also separately either during 1) mixed meal solution (MMS), 2) GIP-, or 3) GLP-1-infusion. Also abdominal subcutaneous and visceral adipose tissue, intestinal and hepatic tissue samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 35 kg/m2
2. Type 2 diabetes mellitus (fasting glucose more than 7 mmol/l)
3. Age: 18-60 years
4. Previous, carefully planned, conservative treatments for obesity have failed

Exclusion Criteria:

1. BMI over 60 kg/m2
2. Weight more than 170 kg
3. Waist circumference > 150 cm
4. Insulin treatment requiring type 2 diabetes mellitus
5. Mental disorder or poor compliance
6. Eating disorder or excessive use of alcohol
7. Active ulcus-disease
8. Pregnancy
9. Past dose of radiation
10. Presence of any ferromagnetic objects that would make MR imaging contraindicated
11. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Inclusion criteria for the control group

1. BMI 18-27 kg/m2
2. Age 18-60 years
3. Fasting plasma glucose less than 6.1 mmol/l
4. Normal glucose tolerance test (OGTT)

Exclusion criteria for the control group

1. Blood pressure > 140/90 mmHg
2. Any chronic disease
3. Mental disorder or poor compliance
4. Any chronic medical defect or injury which hinder/interfere everyday life
5. Eating disorder or excessive use of alcohol
6. Pregnancy
7. Past dose of radiation
8. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results
9. Presence of any ferromagnetic objects that would make MR imaging contraindicated
10. Smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Splanchnic blood flow | 24 months
  Flow is measured using radiowater H2O and PET

SECONDARY OUTCOMES:
GIP and GLP-1 blood concetrations | 24 months
  Blood concentrations are measured from samples

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, Prof, Principal Investigator — PET centre, Turku
Locations (1):
- Turku univercity hospital, PET center, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saari T, Koffert J, Honka H, Kauhanen S, U-Din M, Wierup N, Lindqvist A, Groop L, Virtanen KA, Nuutila P. Obesity-associated Blunted Subcutaneous Adipose Tissue Blood Flow After Meal Improves After Bariatric Surgery. J Clin Endocrinol Metab. 2022 Jun 16;107(7):1930-1938. doi: 10.1210/clinem/dgac191. PMID 35363252
- [Derived] Honka H, Koffert J, Kauhanen S, Teuho J, Hurme S, Mari A, Lindqvist A, Wierup N, Groop L, Nuutila P. Bariatric Surgery Enhances Splanchnic Vascular Responses in Patients With Type 2 Diabetes. Diabetes. 2017 Apr;66(4):880-885. doi: 10.2337/db16-0762. Epub 2017 Jan 17. PMID 28096259